CLINICAL TRIAL: NCT00012519
Title: A Phase I/II Trial of Ritonavir and Indinavir in Children Failing Other Antiretroviral Therapy
Brief Title: Ritonavir and Indinavir in Children Failing Other Anti-HIV Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1013; 10191 (Registry Identifier: DAIDS ES); ACTG P1013; PACTG P1013
Record Dates: First submitted 2001-03-10; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Indinavir; Anti-HIV Agents; Viral Load; Pharmacokinetics; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir

INTERVENTIONS:
Drug: indinavir sulfate
Drug: ritonavir

SUMMARY:
Both ritonavir (RTV) and indinavir (IDV) are approved by the FDA to treat HIV, but IDV has not been approved for use in children and the doses for the combination of the two drugs has not been studied in children. The purpose of this study is to find a combination of RTV and IDV that is safe, well tolerated, and produces drug levels in the blood of children that are comparable to effective drug levels in the blood of adults. The effectiveness of the drug combination in decreasing the amount of virus in the body will also be studied. The children enrolled in this study will have high HIV viral loads despite taking anti-HIV drugs.

DETAILED DESCRIPTION:
Combination regimens of RTV and IDV in adults offer the benefit of two potent antiretroviral agents, convenience of twice-daily dosing, unrestricted timing of meals, and fewer renal complications. There are limited, largely anecdotal data from children suggesting that initial virologic response can also be attained in children given IDV with RTV, but there are not sufficient pharmacokinetic data to define appropriate dose regimens. This study will evaluate the clinical feasibility of a combination RTV and IDV regimen for children.

Patients will be stratified on the basis of age/Tanner stage and ability to swallow intact capsules. Patients will be randomized to either Balanced Dose or Low Dose RTV treatment arms. Patients in the Balanced Dose Arm will receive RTV and IDV in approximately equal doses. The Low Dose RTV Arm will receive a dosing ratio of RTV:IDV of approximately 1:3. Patients will have scheduled study visits every 4 weeks for 6 months, then every 3 months for approximately 18 months. Study visits will consist of a medical history, physical exam, and blood and urine tests. Patients will have intensive pharmacokinetic analysis at Week 4 (or 2 weeks after a stable dose of study drugs has been reached) and Week 16. Study visits that include pharmacokinetic analysis will last 9 to 13 hours.

At each study visit, patients will be closely assessed for drug toxicity and virologic response. At the end of the study, patients with good virologic response and no evidence of toxicity may choose to enter a 48 week extension phase and continue taking the combination regimen.

ELIGIBILITY:
Inclusion Criteria

* HIV infection
* HIV RNA levels > 10,000 copies/ml within 30 days prior to study entry
* Anti-HIV drug therapy failure while on the same anti-HIV drugs for more than 16 weeks
* Body size above a certain limit (body surface area > 0.48 m2)
* Acceptable methods of contraception
* Consent of parent or legal guardian

Exclusion Criteria

* Unable to determine HIV genotypic resistance
* HIV resistant to IDV or RTV at study screening
* Previously received IDV and RTV at the same time
* Need treatment with any medication prohibited by the study
* Glucocorticoids for more than 14 days at study entry
* Cancer requiring chemotherapy
* Drugs affecting the immune system, other than IVIG, within 3 months of study entry
* Certain abnormal laboratory results at study entry
* Pregnant or breast-feeding
* Unable to be followed at a PACTG center during the trial

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Chadwick, Study Chair; Ram Yogev, Study Chair; Stephen Pelton, Study Chair; Elaine Abrams, Study Chair
Locations (12):
- United States (11):
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida College of Medicine-Dept of Peds, Div. of Immunology, Infectious Diseases & Allergy, Gainesville, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Metropolitan Hosp. Ctr., New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
  - VCU Health Systems, Dept. of Peds, Richmond, Virginia
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Saah AJ, Winchell GA, Nessly ML, Seniuk MA, Rhodes RR, Deutsch PJ. Pharmacokinetic profile and tolerability of indinavir-ritonavir combinations in healthy volunteers. Antimicrob Agents Chemother. 2001 Oct;45(10):2710-5. doi: 10.1128/AAC.45.10.2710-2715.2001. PMID 11557459
- [Background] van Rossum AM, de Groot R, Hartwig NG, Weemaes CM, Head S, Burger DM. Pharmacokinetics of indinavir and low-dose ritonavir in children with HIV-1 infection. AIDS. 2000 Sep 29;14(14):2209-10. doi: 10.1097/00002030-200009290-00022. No abstract available. PMID 11061667
- [Background] Chadwick EG, Rodman JH, Samson P, Fenton T, Abrams EJ, Nowak B, Pelton SI, Lavoie S, Knapp K, Bambji M, Yogev R, PACTG 1013 Team. Antiviral Activity, Tolerance and Pharmacokinetics of Indinavir with Two Doses of Ritonavir as Salvage Therapy in Children. 10th Conference on Retroviruses and Oppurtunistic Infections. Feb 2003. Abstract 875.